CLINICAL TRIAL: NCT04400201
Title: A Phase III Clinical Study Evaluating the Efficacy and Safety of Remimazolam Tosilate Compared to Propofol in Patients Undergoing Bronchoscopy
Brief Title: A Clinical Study of Remimazolam Tosilate in Patients Undergoing Bronchoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HR-RMZL-Ⅲ-FB
Record Dates: First submitted 2020-05-14; First posted 2020-05-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2020-05

CONDITIONS: Sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Tosilate (Experimental)
  Interventions: Drug: Remimazolam Tosilate
- Propofol (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam Tosilate — Intravenous injection at a dose of 0.3mg/kg for sedation induction and continuous intravenous infusion at an initiative dose of 1 mg/kg/h for sedation maintenance.
  Arms: Remimazolam Tosilate
Drug: Propofol — Intravenous injection at a dose of 1.5~2.5mg/kg for sedation induction and continuous intravenous infusion at the dose of 0~12 mg/kg/h for sedation maintenance
  Arms: Propofol

SUMMARY:
A multicenter, randomized, single-blind, active controlled, parallel group study comparing remimazolam tosilate to propofol in patients undergoing bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. 18~80 years, female or male
2. Patients scheduled for an bronchoscopy procedure
3. 18 kg/m2<BMI<30kg/m2
4. Patients understand clearly and participate in the study voluntarily, and sign the informed consent

Exclusion Criteria:

1. Patients scheduled for emergency surgery
2. Patients with a history of drug abuse and / or alcohol abuse 2 years prior to the screening period
3. One or more of the laboratory findings fall out of the limitations for this study(platelet,hemoglobin,aspartate aminotransferase,etc.);
4. Pregnant women or those in lactation period
5. Allergic to drugs used in the study
6. Patients have participated in other clinical trial within the 3 months prior to randomization
7. Any patient judged by the Principal Investigator (PI) or Sub-Investigator to be inappropriate for the subject for any other reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of participants who experienced successful sedation in undergoing bronchoscopy in each group | From the onset of administration of the study drug to removal of bronchoscope on Day 1 of treatment

SECONDARY OUTCOMES:
Time from start of investigational medicinal product administration to loss of consciousness | From the onset of administration of the study drug to unconsciousness on Day 1 of treatment
Time from stop of investigational medicinal product to MOAA/S Score=5 | From the last dose of study drug until the patient has recovered to fully alert on Day 1 of treatment
Time from stop of investigational medicinal product to Aldrete Score≥9 | From the end of administration of the study drug until the patient reaches the modified Aldrete's system score of ≥9 points on Day 1 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peking Union Medical College Hospital, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China